CLINICAL TRIAL: NCT07214389
Title: Research to Foster an Opioid Use Disorder Treatment System Patients Can Count On: Project 2 - Producing Outcome Measures for OTP Quality Improvement
Brief Title: PRoducing Outcome Measures for OTP Quality Improvement
Acronym: PROMOTE-QI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: University of California, Los Angeles (Other); BayMark Health Services (Unknown); Los Angeles County Department of Public Health - Substance Abuse Prevention and Control (SAPC) (Unknown); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Tami Mark, Distinguished Fellow, Health Policy, RTI International
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RTI-HEAL-OTP-P2; RM1DA059375 (NIH)
Record Dates: First submitted 2025-10-07; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Opioid Use Disorder
Keywords: Opioid Treatment Programs (OTPs); Methadone; Buprenorphine; Quality Improvement (QI); Treatment Retention; Addiction Services; Implementation Science
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Quality Improvement

STUDY DESIGN:
Intervention Model Description: Parallel-group, cluster-randomized trial at the opioid treatment program (OTP) level. Forty-five BayMark OTPs (~15 per arm) are randomized 1:1:1 to: (1) quality measures + QI toolkit; (2) quality measures + QI toolkit + external QI facilitation (NIATx); or (3) usual care. Patients are not individually assigned; outcomes are derived from routinely collected EHR and Medicaid claims. Enrollment reflects the expected number of adult MOUD initiations during the 12-month post-implementation window across participating sites (~100 per site; total ≈ 4,500). Open-label; analyses account for clustering at the OTP level.
Masking Description: This is an open-label, cluster-randomized implementation trial. OTPs, care providers, and investigators will be aware of arm assignment. Masking is not feasible because the interventions-provision of clinic-level quality measures and a QI toolkit, with or without external QI facilitation-are organizational changes visible to staff. Patient outcomes are obtained from EHR and Medicaid claims; the central analytic team may be masked to arm labels when feasible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 - Title: Quality Measures + QI Toolkit (Experimental): OTPs in this arm receive clinic-level quality measures (claims-based, case-mix-adjusted retention/outcome measures with benchmarks and peer comparisons) plus a self-guided QI toolkit (evidence summaries, change packages, templates, and examples) to support retention-focused practice changes. No external facilitation is provided
  Interventions: Behavioral: Quality Measures (Audit and Feedback); Behavioral: Quality Improvement (QI) Toolkit
- Arm 2 - Title: Quality Measures + QI Toolkit + External QI Facilitation (Experimental): OTPs receive the quality measures and QI toolkit as in Arm 1 plus structured external QI facilitation based on the NIATx model. Facilitators coach an OTP change team, review data, and guide PDSA cycles to implement retention-focused improvements
  Interventions: Behavioral: Quality Measures (Audit and Feedback); Behavioral: Quality Improvement (QI) Toolkit; Behavioral: External QI Facilitation
- Arm 3 - Title: No Intervention: Usual Care (No Intervention): OTPs continue usual practice without access to the quality measures or QI toolkit and with no external facilitation during the study. Outcomes are assessed from EHR and Medicaid claims.

INTERVENTIONS:
Behavioral: Quality Measures (Audit and Feedback) — Clinic-level reports/dashboards providing case-mix-adjusted retention and outcome measures with benchmarks and peer comparisons, derived from EHR and Medicaid claims; delivered periodically to guide quality improvement.
  Arms: Arm 1 - Title: Quality Measures + QI Toolkit; Arm 2 - Title: Quality Measures + QI Toolkit + External QI Facilitation
Behavioral: Quality Improvement (QI) Toolkit — A self-guided QI toolkit for OTPs with step-by-step change packages, PDSA templates, training materials, and case examples to improve retention. Provided together with the quality measures in Arms 1-2; designed for use without external facilitation.
  Arms: Arm 1 - Title: Quality Measures + QI Toolkit; Arm 2 - Title: Quality Measures + QI Toolkit + External QI Facilitation
Behavioral: External QI Facilitation — Structured facilitation based on the NIATx model. Facilitators provide training, coaching, and feedback to an OTP change team, using the measures and toolkit to guide retention-focused QI.
  Arms: Arm 2 - Title: Quality Measures + QI Toolkit + External QI Facilitation

SUMMARY:
This study tests ways to help opioid treatment programs (OTPs) keep patients in care. Staying on methadone or buprenorphine is linked to better outcomes, yet many people leave treatment early. The project will compare two approaches that provide clinics with retention/outcome quality measures and a quality-improvement (QI) toolkit-either alone or with added facilitation-against usual care.

Forty-five BayMark OTPs in multiple states will be randomly assigned to one of three groups: (1) quality measures + QI toolkit; (2) quality measures + QI toolkit + external QI facilitation; or (3) usual care.

The primary outcome is 90-day retention in treatment, measured from OTP electronic health records and Medicaid claims. Secondary outcomes include emergency department visits, hospitalizations, overdoses, and mortality. Findings will identify practical, scalable strategies to improve patient retention in OTPs.

DETAILED DESCRIPTION:
This cluster-randomized trial is part of an NIH/NIDA-funded program to advance quality measurement and management for opioid treatment programs (OTPs). PROMOTE-QI (Project 2) tests whether providing OTPs with retention/outcome quality measures and a quality-improvement (QI) toolkit, with or without additional QI facilitation, improves patient retention compared with usual care. The study is conducted in partnership with BayMark Health Services and academic/industry collaborators.

Design and setting. Forty-five BayMark OTPs in multiple states will be randomized in equal groups to three arms (≈15 sites/arm) in a parallel-group cluster design. We anticipate ~4,500 adult MOUD initiations across the 45 sites during the 12-month post-implementation observation window. Patients are not individually assigned; outcomes are derived from EHR and Medicaid claims.

Interventions. Arm 1: Quality measures + QI toolkit. Sites receive claims-based, case-mix-adjusted retention and outcome quality measures with benchmarks, plus a toolkit (evidence summaries, case studies, and "how-to" materials) to guide retention-focused QI efforts, delivered via a secure portal.

Arm 2: Quality measures + QI toolkit + QI facilitation (NIATx). Sites receive all Arm-1 components plus structured NIATx facilitation, including establishing a change team and running Plan-Do-Study-Act (PDSA) cycles to implement and test retention strategies.

Arm 3: Usual care. Sites continue existing practices; at study end they will be offered the quality-measure portal and toolkit.

Primary and secondary outcomes. The primary endpoint is the OTP's 90-day treatment retention rate. Secondary endpoints are the OTP's 90-day retention rate of medications to treat OUD, the percentage of the OTP's patients with an ED visit or hospitalization for a substance use disorder (SUD), and the percentage with an ED visit or hospitalization for any cause.

Data sources and analysis. Outcomes will be drawn from BayMark electronic health records (EHR) and Medicaid T-MSIS claims. Analyses use generalized linear mixed models that account for clustering at the OTP level; retention/discontinuation rules (e.g., ≥31-day gap) follow the study's measurement specifications.

Implementation outcomes. The study will document strategies adopted, barriers/facilitators, and costs of QI facilitation via surveys/interviews and cost tracking.

Rationale. Prior work shows audit-and-feedback is more effective when paired with actionable guidance; the trial therefore compares quality measures + toolkit with and without facilitation to determine the incremental benefit of NIATx support.

ELIGIBILITY:
Only BayMark OTPs are eligible for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4500 (Estimated)
Dates: Start 2025-10-03 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
OTP's 90-day treatment retention rate | 90 days after treatment initiation (episodes initiating within the 12 months after intervention launch)
  The primary endpoint in the quantitative analyses will be the OTP's 90-day treatment retention rate.

SECONDARY OUTCOMES:
OTP's 90-day retention rate of medications to treat OUD | 90 days after treatment initiation
  The secondary endpoint in the quantitative analysis will be the OTP's 90-day retention rate of medications to treat opioid use disorder.
ED visit or hospitalization for a substance use disorder (SUD) | Within 12 months after treatment initiation (claims-based outcome window)
  the percentage of the OTP's patients who had an emergency department (ED) visit or were hospitalized for a substance use disorder (SUD)
ED visit or hospitalization for any cause | Within 12 months after treatment initiation (claims-based outcome window)
  the percentage of the OTP's patients who had an ED visit or were hospitalized for any cause

CONTACTS AND LOCATIONS:
Overall Officials: Tami L Mark, PhD, Principal Investigator — RTI International
Locations (1):
- RTI International, Research Triangle Park, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study relies on de-identified Medicaid claims and electronic health records obtained through data use agreements, as well as site-level information from opioid treatment programs (OTPs). These data are protected by federal and state privacy regulations and cannot be shared at the participant level. Only aggregated results will be disseminated.